CLINICAL TRIAL: NCT00667888
Title: A Phase III Intensity Radiotherapy Dose Escalation for Prostate Cancer Using Hypofractionation
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID00-381; NCI-2010-01456 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radiation; Radiotherapy; Intensity Modulated Radiotherapy; IMRT; Hypofractionated Intensity Modulated Radiotherapy; HIMRT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensity Modulated Radiotherapy (IMRT) (Active Comparator): A total dose of 75.6 Gy will be delivered in 42 fractions to the planning target volume (PTV).
  Interventions: Radiation: Conventional Fractionated Intensity Modulated Radiotherapy
- Hypofractionated Intensity Modulated Radiotherapy (HIMRT) (Experimental): A total dose of 72 Gy will be delivered in 30 fractions to the PTV.
  Interventions: Radiation: Hypofractionated Intensity Modulated Radiotherapy

INTERVENTIONS:
Radiation: Conventional Fractionated Intensity Modulated Radiotherapy — A total dose of 75.6 Gy will be delivered in 42 fractions to the planning target volume (PTV).
  Other Names: IMRT
  Arms: Intensity Modulated Radiotherapy (IMRT)
Radiation: Hypofractionated Intensity Modulated Radiotherapy — A total dose of 72 Gy will be delivered in 30 fractions to the PTV.
  Other Names: HIMRT
  Arms: Hypofractionated Intensity Modulated Radiotherapy (HIMRT)

SUMMARY:
The goal of this clinical research study is to compare using external beam radiotherapy with intensity modulated beams for fewer days at a higher dose per day to the same type of therapy for more days at a lower dose per day in the treatment of prostate cancer. The safety of these treatments will also be studied and compared.

DETAILED DESCRIPTION:
Patients in this study will be randomly picked (as in the toss of a coin) to be in one of two treatment groups. There is an equal chance of being in either group.

Patients in Group 1 will be treated with intensity modulated radiotherapy (IMRT). These patients will receive 42 treatments, 5 days per week, over 8.5 weeks. This method has become the standard treatment at M.D. Anderson Cancer Center.

Patients in Group 2 will also be treated with IMRT. However, these patients will only receive 30 treatments, 5 days per week, over 6 weeks. The dose per day for Group 2 patients is higher than for Group 1 and has the possibility of killing more tumor cells.

Each external beam treatment requires about 10-20 minutes. However, patients can expect to spend 20 - 30 minutes on the treatment table because imaging measurements of prostate position will be done before each treatment. The total time in the radiation department each treatment day will be about an hour.

After the radiotherapy is completed, patients will have a PSA blood test every 3 months for 2 years, then every 6 months for Years 3 - 5, then annually. They will be examined every 6 months during the first 2 years beginning 3 months after the completion of treatment, then annually. A needle biopsy of the prostate will be performed if these tests suggest recurrence.

This is an investigational study. 225 patients will take part in this study. This study will take place at M. D. Anderson and possibly some affiliated hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proof of adenocarcinoma of the prostate.
2. Bone scan (If PSA >10 ng/ml or T3 disease) within 3 months of starting androgen ablation or signing protocol consent if no androgen ablation.
3. CT-scan of pelvis (If Stage T3 disease) within 3 months of starting androgen ablation or signing protocol consent if no androgen ablation.
4. Suitable medical condition; Zubrod <2.
5. Pretreatment PSA </=20 ng/ml. If PSA <4, must have Gleason greater than or equal to 7 and/or Stage T2b-T2c. PSA within 30 days of signing protocol consent. If neoadjuvant androgen ablation has been given, then the preandrogen ablation PSA should be used for stratification.
6. Clinical (palpable) Stage T1b - T3b disease (1992 AJCC staging system).
7. While a transrectal ultrasound will be obtained before treatment, the staging will not be based on these findings. If palpable T3 disease is present, then must have Gleason score <8 and pretreatment PSA less than or equal to 10 ng/ml
8. Gleason score <10.
9. If Gleason score 8 or 9, then must have stage T1/T2 disease and pretreatment PSA less than or equal to 10 ng/ml.
10. The patient must be able to understand the protocol and adhere to follow-up at 6-month intervals for the first 2 years and at yearly intervals thereafter.
11. Informed consent must be given.
12. Patients randomized to Arm 1 may also participate in protocol 2004-0428.

Exclusion Criteria:

1. Prior pelvic radiotherapy.
2. Greater than 4 months of prior hormone ablation therapy.
3. Prior or planned radical prostate surgery.
4. Clinical, radiographic or pathologic evidence of nodal or distant metastatic disease.
5. Concurrent, active malignancy, other than nonmetastatic skin cancer or early stage -chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma). If a prior malignancy is in remission for greater than or equal to 5 yr then the patient is eligible.
6. Zubrod status greater than or equal to 2.
7. Pretreatment PSA >20 ng/ml.
8. Gleason score of 10.
9. Palpable stage T3c (seminal vesicle involvement) or T4 disease.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2001-01-03 (Actual); Primary Completion 2015-10-12 (Actual); Study Completion 2021-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A. Kuban, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hassanzadeh C, Kuban D, Pasyar S, Bassett R, Troncoso P, Ansari M, Schlembach P, McGuire S, Nguyen Q, Frank S, Mok H, Mohamad O, Park R, Tang C, Du W, Kudchadker R, Choi S, Hoffman K. Hypofractionated, Dose-Escalated Radiation Versus Conventionally Fractionated Radiation for Localized Prostate Cancer: Long-Term Update of a Phase III, Prospective, Randomized Controlled Trial. J Clin Oncol. 2025 Jun 20;43(18):2044-2048. doi: 10.1200/JCO-24-02057. Epub 2025 May 14. PMID 40367400
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients referred for radiotherapy with histologically proven adenocarcinoma of the prostate with clinical stage T1b-T3b disease and without clinical radiographic evidence of metastasis from 2001-2010.
Pre-assignment Details: 225 patient enrolled on the trial, 222 patients met criteria and participated to be randomized on trial. 203 patients were deemed evaluable.
Groups:
- Arm 1: (CIMRT) Conventional Radiotherapy: Patients' radiotherapy plan includes 75.6 Gy in 1.8-Gy fractions delivered over 8.4 weeks
- Arm 2: (HIMRT) Hypofractionated Radiotherapy: Patients' radiotherapy plan includes 72 Gy in 2.4 Gy fractions delivered over 6 weeks
Period: Overall Study
Arm/Group | Arm 1: (CIMRT) Conventional Radiotherapy | Arm 2: (HIMRT) Hypofractionated Radiotherapy
Started | 111 | 111
Completed | 101 | 102
Not Completed | 10 | 9
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Proceed with other treatment | 3 | 3
Not completed — Ineligible after SIM | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: (CIMRT) Conventional Radiotherapy | Arm 2: (HIMRT) Hypofractionated Radiotherapy | Total
Number analyzed (Participants) | 111 | 111 | 222
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 38 | 87
  >=65 years | 62 | 73 | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 111 | 111 | 222
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 100 | 104 | 204
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 13 | 31
  White | 85 | 93 | 178
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 111 | 111 | 222

OUTCOME MEASURES:

1. Primary Outcome: Conventional Radiotherapy (CIMRT) Versus Hypofractionated Radiotherapy (HIMRT)
Description: To determine the progression of the number of participants who failed treatment after receiving (CIMRT) versus (HIMRT). PSA measured on (CIMRT) and (HIMRT) for each participant on both arms. Failure was defined as Prostate-specific antigen (PSA) failure using the Phoenix definition of nadir plus 2 ng/ml, or initiation of salvage therapy.
Time Frame: 8.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: (CIMRT) Conventional Radiotherapy | Arm 2: (HIMRT) Hypofractionated Radiotherapy
Number analyzed (Participants) | 101 | 102
Participants | 21 | 10

ADVERSE EVENTS:
Time Frame: 8.5 years
Arm/Group | Arm 1: (CIMRT) Conventional Radiotherapy | Arm 2: (HIMRT) Hypofractionated Radiotherapy
All-Cause Mortality (participants affected / at risk) | 1/101 | 1/102
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/102
Other Adverse Events (participants affected / at risk) | 56/101 | 79/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: (CIMRT) Conventional Radiotherapy (N=101) | Arm 2: (HIMRT) Hypofractionated Radiotherapy (N=102)
Hematuria (Renal and urinary disorders) | 5 | 7
Discomfort (Renal and urinary disorders) | 2 | 3
Frequency (Renal and urinary disorders) | 17 | 12
Incontinence (Renal and urinary disorders) | 1 | 5
Urgency,Retention, Hesitancy/weak stream, Strictured (Renal and urinary disorders) | 5 | 12
Frequency (Gastrointestinal disorders) | 1 | 2
Discomfort (Gastrointestinal disorders) | 4 | 2
Urgency,Retention, Hesitancy/weak stream, Strictured (Gastrointestinal disorders) | 2 | 3
Bleeding (Gastrointestinal disorders) | 19 | 32
Incontinence (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes